CLINICAL TRIAL: NCT01172405
Title: A Clinical Multicenter, Phase III, Randomized, Double-blind, Prospective and Comparative Trial to Evaluate the Efficacy and Safety of the Combination of Ibuprofen + Caffeine in the Treatment of Headache Attacks, Compared to Ibuprofen Alone.
Brief Title: Efficacy and Safety Study to Compare Ibuprofen + Caffeine With Ibuprofen Alone in the Treatment of Headache
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mantecorp Industria Quimica e Farmaceutica Ltd. (Industry)
Responsible Party: Celso Pereira Sustovich, Medical Director, Mantecorp Indústria Química e Farmacêutica Ltda.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IBU-CAF-01/09
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2010-07

CONDITIONS: Headache
Keywords: Headache; Migraine; Ibuprofen; Caffeine
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Ibuprofen; Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibuprofen + Caffeine (Experimental): 72 patients treated with one or two tablets of ibuprofen 400 mg + caffeine 200 mg when presenting headache.
  Interventions: Drug: Ibuprofen plus caffeine
- Ibuprofen (Active Comparator): 72 patients treated with one or two tablets of ibuprofen 400 mg when presenting headache.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen plus caffeine — One or two tablets of ibuprofen 400 mg + caffeine 200 mg when presenting headache.
  Arms: Ibuprofen + Caffeine
Drug: Ibuprofen — One or two tablets of ibuprofen 400 mg when presenting headache.
  Other Names: DALSY
  Arms: Ibuprofen

SUMMARY:
Based on established therapeutic effect of ibuprofen in the treatment of headache attacks, and the action of caffeine in promoting better results when combined with treatments of first choice in the treatment of headache, this study is designed to:

* evaluate the efficacy of therapy with ibuprofen + caffeine in headache patients compared to ibuprofen alone;
* evaluate the tolerability of the association ibuprofen + caffeine compared to ibuprofen alone.

The hypothesis is that the association is superior to treatment with ibuprofen alone in terms of efficacy, while maintaining good tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ability to read, understand and sign the IC;
* Patients with symptoms of frequent episodic tension headache, mild to moderate;
* Patients with symptoms of migraine with or without aura, of mild to moderate intensity;
* Patients who have had between two and five headache attacks in the last 30 days;
* Patients who accept the condition of ingesting less than three cups of coffee per day and / or reduce the intake of any beverage that contains caffeine;
* Patients who accept the condition not to drink any beverage that contains caffeine for 24 hours after drug administration.
* Patients able to understand and maintain the clinical protocol.
* Patients who started or changed prophylactic treatment for headache 30 days before inclusion.
* Female patients of childbearing age must agree to undergo pregnancy testing through urine.

Exclusion Criteria:

* Patients in whom headache began after 50 years of age;
* Patients with strong or disabling headaches;
* Patients with chronic daily headaches lasting up to 72 h or with cluster headaches not responsive to common analgesics;
* Patients with headaches occurring in 15 or more days per month;
* Patients with secondary headaches;
* Patients who overuse analgesics (acetylsalicylic acid up to 300 mg / day) or NSAIDs;
* Known hypersensitivity to components of both formulations of the drug test as the comparison;
* Known hepatic or renal diseases;
* Patients who are pregnant or intend to become pregnant or lactating;
* Patients with severe concomitant systemic diseases such as cancer, diabetes, congenital or acquired heart diseases, hematological diseases, convulsive disorders, autoimmune diseases, renal failure, severe infections, hormonal disorders, pulmonary disorders and peptic diseases;
* History of alcoholism or substance abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of study treatment compared with control to relieve headache symptoms. | 4 weeks
  The evaluation of efficacy will be determined based on comparison of the intensity of headache before and after initiation of treatment, using the Functional Disabling Scale. The opinion of the investigator will be established based on the Likert scale and duration of symptoms after the treatment will be checked as a measure of comparison between treatments in the study.

SECONDARY OUTCOMES:
Tolerability of study treatment compared with control to relieve headache symptoms. | 4 weeks
  Tolerability will be assessed by the investigator through the number of adverse events definitely related to study medication. This relationship will be defined by applying the Naranjo algorithm.